CLINICAL TRIAL: NCT06983691
Title: Evaluating a Patient Navigation Program to Improve Therapy Management for HER2+ Metastatic Breast Cancer Patients Treated With Tucatinib
Brief Title: Patient Navigation for HER2+ Metastatic Breast Cancer Patients Treated With Tucatinib
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro00117920
Record Dates: First submitted 2025-05-14; First posted 2025-05-21 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: HER2+ Metastatic Breast Cancer (MBC)
Keywords: Patient Navigation
MeSH Terms: interventions — Patient Navigation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient Navigation Program (Experimental): The patient navigation program will integrate 1) education to enhance understanding of the treatment regimen, follow-up care, and the importance of adherence, 2) symptom management and adherence strategies, and 3) skills and resources to enhance women's symptom coping and self-management abilities.
  Interventions: Behavioral: Patient Navigation Program

INTERVENTIONS:
Behavioral: Patient Navigation Program — The patient navigation program will integrate 1) education to enhance understanding of the treatment regimen, follow-up care, and the importance of adherence, 2) symptom management and adherence strategies, and 3) skills and resources to enhance women's symptom coping and self-management abilities.

SUMMARY:
The goal of this study is to test a novel nurse-delivered patient navigation program for women with HER2+ metastatic breast cancer (mBC) receiving tucatinib, trastuzumab, and capecitabine. The program will focus on enhancing understanding of the treatment regimen, managing symptoms and adherence, and improving coping and self-management skills. If successful, the program could be integrated into clinical care to better support mBC patients. The main question the study aims to answer is: is the patient navigation program feasible and acceptable for mBC patients?

Participants will receive patient navigation sessions over about 12 weeks. Participants will also complete study assessments via electronic survey at baseline and at about 3, 6, 9, and 12 weeks after enrollment, with the last assessment occurring after completion of the patient navigation program sessions. Participants will also complete a post-program exit interview.

ELIGIBILITY:
Inclusion Criteria:

* female (sex assigned at birth);
* ≥18 years of age at enrollment;
* diagnosed with HER2+ metastatic breast cancer (mBC);
* receiving treatment with tucatinib combined with capecitabine and trastuzumab;
* able to speak and read English

Exclusion Criteria:

* visual or hearing impairment;
* severe cognitive impairment;
* severe mental illness interfering with ability to participate

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Number of participants enrolled | 9 months
  Feasibility will be assessed by examining pilot study enrollment.
Percentage of participants completing 3 sessions | 12 weeks
  Feasibility will be assessed by examining retention (>80% completing 3 sessions).
Percentage of participants using program strategies | 12 weeks
  Feasibility will be assessed by examining use of program strategies (≥75% reporting use of program skills and strategies).
Treatment Acceptability Questionnaire (TAQ) score | 12 weeks
  Acceptability will be assessed using the Treatment Acceptability Questionnaire (TAQ). The program will be considered acceptable if >80% of participants rate the program as >5 out of 7 on the TAQ. A higher score indicates greater acceptability.
Client Satisfaction Questionnaire (CSQ) score | 12 weeks
  Acceptability will be assessed using the Client Satisfaction Questionnaire (CSQ). The program will be considered acceptable if >80% of participants rate the program as >3 out of 4 on the CSQ. A higher score indicates greater acceptability.

OTHER OUTCOMES:
Change in percentage of correct items on a knowledge assessment | Baseline to 12 weeks
  Knowledge will be assessed using an item pool developed for the study. Each participant will complete 10 items based on the education they received. Knowledge will be calculated as the percent of correct items.
Change in adherence as measured by number of participants with discontinuation | Baseline to 12 weeks
  Adherence will be measured for each drug in the regimen as discontinuation (yes/no).
Change in adherence as measured by Voils' medication adherence self-report measure | Baseline to 12 weeks
  For oral medications (i.e., tucatinib, capecitabine), medication taking behaviors (implementation adherence) will be measured using the Voils' medication adherence self-report measure which assesses the extent of (3 items) and reasons (18 items) for non-adherence.
Change in symptom severity as measured by the MD Anderson Symptom Inventory (MDASI) | Baseline to 12 weeks
  The MDASI assesses the severity of symptoms at their worst in the last 24 hours on a 0-10 numerical rating scale, with 0 being "not present" and 10 being "as bad as you can imagine."
Change in symptom interference as measured by the MD Anderson Symptom Inventory (MDASI) | Baseline to 12 weeks
  The MDASI measures how much the symptoms have interfered with six daily activities: general activity, mood, work, relations with others, walking, and enjoyment of life. Interference is rated on a 0-10 numerical rating scale, 0 being "did not interfere" and 10 being "interfered completely."
Change in the impact of hand-foot syndrome (HFS) on quality of life as measured by the Hand-Foot Syndrome Quality of Life Scale (HFS-14) | Baseline to 12 weeks
  The HFS-14 score is calculated by summing the scores of all items and was adjusted to 100 by applying a rule of three. HFS-14 scores are in the range of 2-100, where a higher score indicates greater quality of life impairment.
Change in anxiety severity as measured by the Patient-Reported Outcomes Measurement Information System (PROMIS) Anxiety 4-item Short-Form | Baseline to 12 weeks
  The PROMIS Anxiety Short Form is scored by summing the individual item scores, with each item rated on a 1-5 Likert scale (never, rarely, sometimes, often, always). The total raw score ranges from 4 to 20, where higher scores indicate greater anxiety severity.
Change in depression severity as measured by the Patient-Reported Outcomes Measurement Information System (PROMIS) Depression 4-item Short-Form | Baseline to 12 weeks
  The PROMIS Depression Short Form is scored by summing the individual item scores, with each item rated on a 1-5 Likert scale (never, rarely, sometimes, often, always). The total raw score ranges from 4 to 20, where higher scores indicate greater depression severity.
Change in quality of life as assessed by the Functional Assessment of Cancer Therapy - Breast (FACT-B) | Baseline to 12 weeks
  Quality of life will be assessed using the Functional Assessment of Cancer Therapy - Breast (FACT-B). The FACT-B total score ranges from 0 to 148, where a higher score indicates better quality of life.
Change in self-efficacy as measured by the Patient-Reported Outcomes Measurement Information System (PROMIS) Self-efficacy for Managing Symptoms 4-item Short Form | Baseline to 12 weeks
  The PROMIS Self-efficacy for Managing Symptoms Short Form is scored by summing the individual item scores, with each item rated on a 1-5 Likert scale (never, rarely, sometimes, often, always). The total raw score ranges from 4 to 20, where higher scores indicate greater self-efficacy.
Change in self-efficacy as measured by the Patient-Reported Outcomes Measurement Information System (PROMIS) Self-efficacy for Managing Chronic Conditions 4-item Short Form | Baseline to 12 weeks
  The PROMIS Self-efficacy for Managing Chronic Conditions Short Form is scored by summing the individual item scores, with each item rated on a 1-5 Likert scale (never, rarely, sometimes, often, always). The total raw score ranges from 4 to 20, where higher scores indicate greater self-efficacy.
Change in patient activation as measured by the Patient Activation Measure (PAM) | Baseline to 12 weeks
  The PAM assesses patients' knowledge, skills, and confidence central to managing their health and health care. Patients rate how much they agree or disagree with each item; raw scores are transformed to a score of 0-100, where a higher score indicates greater activation.

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Shelby, PhD, Principal Investigator — Duke University

IPD SHARING:
Plan to Share IPD: No